CLINICAL TRIAL: NCT01940354
Title: A Prospective, Randomized, Controlled Comparison of First Attempt Success Between the AccuCath Intravenous System With Retractable Coiled Tip Guide Wire and Conventional Peripheral Intravenous Catheters With Interventional Radiology Nurses
Brief Title: Comparison of AccuCath IV Catheter and Conventional IV Catheter in Interventional Radiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VPW-STP-00003
Record Dates: First submitted 2013-09-03; First posted 2013-09-12 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Vascular Access Complications
Keywords: IV Catheter comparison; AccuCath versus Conventional IV Catheters; IV Catheter Study; IV Catheter User Preference Comparison; First Attempt Success Rate for IV Catheters; AccuCath Device Performance; Patient Satisfaction with IV Catheters; Clinician Satisfaction with AccuCath Device Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vascular access via study device (Experimental): AccuCath IV Catheter System will be used for IV therapy during interventional radiology procedure. Intervention includes vascular access, fluid infusion, and blood sample removal.
  Interventions: Device: AccuCath IV Catheter System
- Vascular access via control device (Active Comparator): Conventional IV Catheter System (current catheter) will be used for IV therapy during interventional radiology procedure. Interventions include vascular access, administration of fluids, and blood sample removal.
  Interventions: Device: Conventional IV Catheter System

INTERVENTIONS:
Device: AccuCath IV Catheter System — Vascular access and indwelling catheter placement via study device for infusion of fluids and removal of blood samples.
  Other Names: Rapid Intravascular Start System (RIVS); AccuCath System
  Arms: Vascular access via study device
Device: Conventional IV Catheter System — Vascular access and indwelling catheter placement via control device for infusion of fluids and removal of blood samples
  Arms: Vascular access via control device

SUMMARY:
The study will test a hypothesis that the AccuCath™ System will have a higher rate of successful first attempt peripheral IV placement and higher clinician and patient satisfaction compared to Conventional IV Catheters.

DETAILED DESCRIPTION:
This study is designed to evaluate user/physician preference as it relates to use of a 510(k) cleared vascular access peripheral IV catheter device compared with peripheral IV conventional needle/catheter devices, in terms of first stick success rates, adverse events and overall user and patient satisfaction. As noted above, the study is designed to formally test the hypothesis that the AccuCath™ System will exhibit superiority in terms of the rate of successful first attempt peripheral IV placement and higher user and patient satisfaction compared to Conventional IV Catheters.

ELIGIBILITY:
* Inclusion Criteria:

  1. Male or female, age > or equal to 18 years or < or equal to 89 years old;
  2. Capable and willing to give informed consent;
  3. English speaking;
  4. Acceptable candidate for an elective, non-emergent peripheral intravenous (PIV) catheter placement as determined by ordering physician;
  5. Admitted to study area.

Exclusion Criteria:

1. Male or female, < 18 years old or > 89 years old;
2. Requirement for emergent IV placement (patient's condition would be compromised if there is a delay in IV placement);
3. Previous venous grafts or surgery at the target vessel access site;
4. Currently involved in other investigational clinical trials (unless permission is granted by other study PI).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott O Trerotola, BA, MD, Principal Investigator — University of Pennsylvania; William Stavropoulos, MD, Principal Investigator — Hosptial of the University of Pennsylvania; Suzanne Sweeney, RN, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from April 2013 - November 2013. Location was Interventional Radiology Department at participating hospital.
Groups:
- Vascular Access Via Study Device: AccuCath IV Catheter System will be used for IV therapy during interventional radiology procedure. Intervention includes vascular access, fluid infusion, and blood sample removal.
  AccuCath IV device: Vascular access and indwelling catheter placement via study device for infusion of fluids and removal of blood samples.
- Vascular Access Via Control Device: Conventional IV Catheter (current catheter) will be used for IV therapy during interventional radiology procedure. Interventions include vascular access, administration of fluids, and blood sample removal.
  Conventional IV catheters: Vascular access and indwelling catheter placement via control device for infusion of fluids and removal of blood samples
Period: Overall Study
Arm/Group | Vascular Access Via Study Device | Vascular Access Via Control Device
Started | 110 | 110
Completed | 106 | 108
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vascular Access Via Study Device | Vascular Access Via Control Device | Total
Number analyzed (Participants) | 110 | 110 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 71 | 152
  >=65 years | 29 | 39 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 34 | 81
  Male | 63 | 76 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 28 | 55
  White | 73 | 70 | 143
  More than one race | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 110 | 110 | 220

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rate With Peripheral IV (PIV) Catheter Placement
Time Frame: Baseline/at catheter placement, PIV placement duration ranges from 3-15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Vascular Access Via Study Device | Vascular Access Via Control Device
Number analyzed (Participants) | 110 | 110
Participants | 84 | 90

2. Secondary Outcome: Patient Satisfaction Upon Successful PIV Placement
Description: Patient Satisfaction was measured at initial PIV placement using a 5 Point Likert Scale: 5 - Very Comfortable, 4 - Somewhat Comfortable, 3 - Neutral, 2- Somewhat Uncomfortable, 1 - Very Uncomfortable
Time Frame: Baseline/at catheter placement; PIV placement duration ranges from 3-15 minutes
Population: The number of patients analyzed in each group differs from the numbers in the Participant Flow due to missing data (n = 6 in Study Device arm and n = 1 in the Control Arm).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vascular Access Via Study Device | Vascular Access Via Control Device
Number analyzed (Participants) | 104 | 109
units on a scale | 3.88 (1.11) | 4.46 (0.95)

3. Secondary Outcome: Clinician Satisfaction Upon Successful PIV Placement
Description: Clinician Satisfaction was measured at initial PIV placement using a 5 Point Likert Scale: "How easy was the AccuCath™ System to use in comparison to the current catheter?" 5 - Easier to Use 4 - Somewhat Easier to Use 3 - Neutral 2 - Somewhat Difficult to Use
  1 - Very Difficult to Use
Time Frame: Baseline/at catheter placement; PIV placement duration ranges from 3-15 minutes
Population: The number of patients analyzed in each group differs from the numbers in the Participant Flow due to missing data (n = 5 in Study Device arm and n = 1 in the Control Arm).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vascular Access Via Study Device | Vascular Access Via Control Device
Number analyzed (Participants) | 105 | 109
units on a scale | 3.27 (1.11) | 3.48 (1.04)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant from post-PIV placement until catheter removal (up to 14 days).
Arm/Group | Vascular Access Via Study Device | Vascular Access Via Control Device
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/110
Other Adverse Events (participants affected / at risk) | 2/110 | 10/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vascular Access Via Study Device (N=110) | Vascular Access Via Control Device (N=110)
Infiltration (Vascular disorders) | 2 (2) | 8 (8)
Hematoma (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No